CLINICAL TRIAL: NCT04367805
Title: Impact of COVID-19 Infection in Patients With Hepatocellular Carcinoma: An Ambispective Study Nestled in the CHIEF Cohort
Brief Title: COVID-19 Infection in Patients With Hepatocellular Carcinoma
Acronym: COVID19-CHIEF
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier-Universitaire Bondy (Unknown); University Hospital, Bordeaux (Other); Centre Hospitalier-Universitaire CLICHY (Unknown); Centre Hospitalier Général CORBEIL-ESSONNE (Unknown); CHU CRETEIL (Unknown); University Hospital, Grenoble (Other); University Hospital, Lille (Other); Hospices Civils de Lyon (Other); Poitiers University Hospital (Other); Rennes University Hospital (Other); University Hospital, Rouen (Other); University Hospital, Toulouse (Other); CHU VILLEJUIF (Unknown); Central Hospital, Nancy, France (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0042
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma; COVID-19
Keywords: Hepatocellular Carcinoma; COVID-19; Coronavirus disease 2019-Incidence
MeSH Terms: conditions — Carcinoma, Hepatocellular; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: nasopharyngeal Covid 19 RT-PCR — nasopharyngeal Covid 19 RT-PCR

SUMMARY:
Since December 2019, a new disease named COVID-19 linked to a new coronavirus, SARS-CoV2 has emerged in China in the city of Wuhan, Hubei province, spreading very quickly to all 5 continents, and responsible for a pandemic. France is the third most affected country in Europe after Italy and Spain. Groups of patients at a higher risk of developing a severe form of COVID-19 have been defined: this include patients with immunosuppressive disease as cancer or patients with advanced cirrhosis of the liver. Coronavirus liver injury had been described with SARS-CoV 1 and MERS-CoV. There is no data on liver damage associated with COVID-19 infection for compensated or decompensated cirrhotic patients. The objectives of this project are to estimate the incidence of COVID-19 in hepatocellular carcinoma population, both hospital and ambulatory, and to study the impact on the frequency of severe forms, the prognosis, but also liver function, and the management of hepatocellular carcinoma, in this context of pandemic

ELIGIBILITY:
Inclusion Criteria:

* Patients with CHC and included in the French national prospective cohort CHIEF
* Hospital and ambulatory patients
* Infection confirmed by COVID-19 defined by a positive nasopharyngeal PCR or if PCR COVID-19 negative : CT showing COVID-19 compatible pneumonia
* Suspected COVID-19 infection, not confirmed by COVID-19 PCR or chest CT, with no other known cause of acute pneumonia.

Exclusion Criteria:

* Patient refusal
* Influenza only, confirmed by a diagnostic test
* Other proven causes of pneumonia and absence of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hepatocellular carcinoma population, both hospital and ambulatory
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of COVID-19 infection in patients with hepatocellular carcinoma in France | 6 months
  Incidence of COVID-19 infection in patients with hepatocellular carcinoma in France

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No